CLINICAL TRIAL: NCT07167329
Title: The BELIEVE-VHL Trial: A Real-world Longitudinal Study on Belzutifan's Effectiveness, Pharmacogenetics, and Pharmacoeconomics in Von Hippel-Lindau (VHL) Syndrome Using the HIF2α Inhibitor Belzutifan
Brief Title: Real-World Effectiveness and Pharmacogenetics of Belzutifan in VHL Syndrome: The BELIEVE-VHL Trial
Acronym: BELIEVE-VHL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: José Claudio Casali da Rocha (Other)
Collaborators: AC Camargo Cancer Center (Other)
Responsible Party: Sponsor-Investigator, José Claudio Casali da Rocha, Head of Department of Oncogenetics, AC Camargo Cancer Center
Organization: AC Camargo Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCamargoCC
Record Dates: First submitted 2025-01-25; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Von Hippel Lindau; Von Hippel Lindau Disease; Von Hippel Lindau-Deficient Clear Cell Renal Cell Carcinoma; Hemangioblastoma (HB) of the Central Nervous System (CNS); PNET; Retinal Angiomatous Proliferation; Pheochromocytoma/Paraganglioma; Endolymphatic Sac Tumor
Keywords: Belzutifan; von Hippel-Lindau; Renal Cell Clear Carcinoma; Hemangioblastoma of Central Nervous System; Pharmacogenetics
MeSH Terms: conditions — von Hippel-Lindau Disease; Hemangioblastoma; Neuroectodermal Tumors, Primitive; Pheochromocytoma; Paraganglioma; Carcinoma, Renal Cell | interventions — belzutifan

STUDY DESIGN:
Intervention Model Description: The BELIEVE-VHL Trial is a prospective cohort study designed to evaluate the effectiveness and adverse effects of belzutifan in 100 patients with von Hippel-Lindau syndrome enrolled in a single intervention arm. The trial is structured as a basket trial, including all VHL-associated tumors, in patients aged 14 years or older and at any disease stage. The intervention consists of oral administration of belzutifan (Welireg) 120 mg once daily in patients with clinically or genetically confirmed VHL who are symptomatic or present with progressive tumors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral Belzutifan (WELIREG™) (Experimental): Patients with von Hippel-Lindau Syndrome presenting with lesions or neoplasms requiring treatment with oral Belzutifan (WELIREG™)
  Interventions: Drug: Belzutifan

INTERVENTIONS:
Drug: Belzutifan — Patients with Von Hippel-Lindau Syndrome presenting with lesions or neoplasms requiring treatment with oral Belzutifan.

SUMMARY:
The BELIEVE-VHL Trial is a prospective real-life study designed to evaluate the therapeutic effects, benefits, and adverse effects of belzutifan, as well as the timing of treatment response and disease progression in patients with von Hippel-Lindau (VHL) syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To evaluate the therapeutic effects, benefits, and adverse effects associated with belzutifan treatment, as well as the timing of treatment response and/or disease progression.

SECONDARY OBJECTIVES

1. To evaluate the association of host intrinsic factors with toxicity and treatment response in a Brazilian cohort of patients with von Hippel-Lindau syndrome treated with belzutifan.
2. To assess hemoglobin and erythropoietin levels during the first six months of treatment, and to document the need for subcutaneous erythropoietin supplementation in patients who develop grade 2-3 anemia, fatigue, or hypoxia.
3. To evaluate the potential impact of erythropoietin supplementation on tumor growth during belzutifan treatment.
4. To assess health-related quality of life and patient perceptions regarding VHL syndrome using validated questionnaires and instruments.
5. To conduct a pharmacoeconomic analysis in the cohort of patients with access to belzutifan, assessing its impact on healthcare costs compared to the natural history of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 14 years.
* Clinical or genetic confirmation of von Hippel-Lindau (VHL) syndrome.
* Presence of measurable or progressive VHL-associated tumors, as defined by RECIST 1.1 or disease-specific imaging criteria.
* ECOG performance status of 0-2.
* Adequate bone marrow, hepatic, and renal function as defined by laboratory reference values.
* Ability to swallow oral medication.
* Provision of written informed consent prior to enrollment.

Exclusion Criteria:

* Age < 14 years.
* Absence of a confirmed diagnosis of von Hippel-Lindau (VHL) syndrome.
* Presence of an active malignancy outside the VHL tumor spectrum within the past 3 years, except for adequately treated basal or squamous cell carcinoma of the skin, cervical carcinoma in situ, or other malignancies considered cured for >2 years.
* Known hypersensitivity or allergic reaction to belzutifan or any excipient in the formulation.
* History of severe or uncontrolled cardiovascular disease, including but not limited to unstable angina, myocardial infarction within the past 6 months, congestive heart failure requiring treatment, or uncontrolled hypertension.
* Active infectious diseases, including HIV, hepatitis B, or hepatitis C.
* Immunosuppressed status, whether due to underlying disease or ongoing therapy.
* History of significant bleeding disorders, including bleeding diathesis, thrombocytopenia, or coagulopathy.
* Radiotherapy administered within 4 weeks prior to study enrollment.
* Major surgical procedure, including for VHL-related tumors, within 4 weeks prior to study enrollment, or immediate need for surgical intervention for tumor management.
* Malabsorption secondary to prior gastrointestinal surgery or active gastrointestinal disease.
* Current use of concomitant medications known to interact with belzutifan and significantly alter its bioavailability.
* Anticipated low adherence to or planned interruption of belzutifan therapy.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective Tumor Response per RECIST 1.1 | From enrollment and initiation of treatment until the earliest of either documented disease progression or death from any cause, with follow-up of up to 104 weeks.
  Evaluation of target lesion size according to RECIST 1.1 criteria at baseline, weeks 12, 24, 52, and annually, up to 104 weeks. Imaging modalities will include MRI for solid tumors, 68Ga-DOTATATE PET for pancreatic neuroendocrine tumors (PNET), and retinal fluorescein angiography (FA) for retinal lesions.
  Unit of Measure: Percentage of participants with objective response.

SECONDARY OUTCOMES:
Incidence of Anemia (per CTCAE v5.0) | Baseline to 104 weeks
  Number of participants developing grade ≥2 anemia during treatment with belzutifan, evaluated according to CTCAE version 5.0.
  Correlate hematologic outcomes with tumor response (RECIST 1.1) and lesion dynamics to identify potential predictive biomarkers.
  Unit of Measure: Percentage of participants.
Mean Hemoglobin Level Over Time | Baseline to 104 weeks.
  Longitudinal change in hemoglobin levels (g/dL) at months 1, 3, 6, 12, and annually thereafter.
  Unit of Measure: g/dL.
Erythropoietin Levels Over Time | Time Frame: Baseline to 104 weeks
  Longitudinal change in endogenous erythropoietin levels (mIU/mL) at months 1, 3, 6, 12, and annually thereafter.
  Unit of Measure: mIU/mL.
Requirement for Erythropoietin Supplementation | Baseline to 104 weeks
  Proportion of participants requiring subcutaneous erythropoietin supplementation for symptomatic or grade ≥3 anemia, including dose, frequency, and duration.
  Unit of Measure: Percentage of participants.
Blood Transfusion Requirement | Baseline to 104 weeks
  Number of participants requiring at least one blood transfusion during treatment with belzutifan.
  Unit of Measure: Percentage of participants.
Patient-Reported Quality of Life (EORTC QLQ-C30) | Baseline to 24 months
  Change in health-related quality of life scores measured by the EORTC QLQ-C30: The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30, version 3.0, at baseline, months 1, 3, 6, 12, and annually thereafter.
  It consists of 28 items evaluating symptom burden and functional status, each scored on a 4-point Likert scale (1 = "Not at all," 2 = "A little," 3 = "Quite a bit," 4 = "Very much"). In addition, two items assess overall health and overall quality of life, each rated on a 7-point scale (1 = "Very poor" to 7 = "Excellent") All treatment modifications-including interruptions, dose reductions, or discontinuations-will be recorded throughout the study.
  Unit of Measure: Score from 0 to 100 (higher score indicates better quality of life).
Pharmacoeconomic Evaluation of Belzutifan Therapy in Individuals with von Hippel-Lindau Syndrome | Retrospective analysis of the 5 years prior to belzutifan initiation and prospective follow-up for up to 2 years after treatment initiation.
  The pharmacoeconomic analysis will be conducted in the same cohort of participants treated with belzutifan. Retrospective data on direct medical costs, expressed in Brazilian Reais (R$), will be collected, including expenses related to medications, surgical procedures, and hospital admissions. Indirect costs, particularly those related to productivity losses, will also be assessed and quantified as a percentage reduction compared with healthy employees or as hours/days lost due to illness or treatment-related absenteeism during the preceding five years. All cost data will be analyzed on a per-patient-per-month (PPPM) basis, stratified by defined time intervals. Cost-effectiveness will be evaluated by comparing healthcare costs before and after belzutifan initiation, accounting for changes in procedure frequency and overall resource utilization. Unit of Measure: Brazilian Reais (R$) per PPPM.

CONTACTS AND LOCATIONS:
Locations (1):
- AC Camargo Cancer Center, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share anonymized clinical and laboratorial data, outcomes, side effects, pharmacogenomic information, and their correlation with treatment. This will enable collaboration with other researchers to combine findings and enhance statistical power.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At any time of the study as the results are analyzed, publicly presented and published
Access Criteria: Data will be shared after Transfer Data Agreement between Principal Investigators and institutions, based on new bilateral approval on Ethics and Research Committees of both involved oncology centers.

REFERENCES:
- [Background] Else T, Jonasch E, Iliopoulos O, Beckermann KE, Narayan V, Maughan BL, Oudard S, Maranchie JK, Iversen AB, Goldberg CM, Fu W, Perini RF, Liu Y, Linehan WM, Srinivasan R. Belzutifan for von Hippel-Lindau Disease: Pancreatic Lesion Population of the Phase 2 LITESPARK-004 Study. Clin Cancer Res. 2024 May 1;30(9):1750-1757. doi: 10.1158/1078-0432.CCR-23-2592. PMID 38393723
- [Background] Eriksson M, Lindstrom B. Validity of Antonovsky's sense of coherence scale: a systematic review. J Epidemiol Community Health. 2005 Jun;59(6):460-6. doi: 10.1136/jech.2003.018085. PMID 15911640
- [Background] Bagattini AM, Camey SA, Miguel SR, Andrade MV, de Souza Noronha KVM, de C Teixeira MA, Lima AF, Santos M, Polanczyk CA, Cruz LN. Electronic Version of the EQ-5D Quality-of-Life Questionnaire: Adaptation to a Brazilian Population Sample. Value Health Reg Issues. 2018 Dec;17:88-93. doi: 10.1016/j.vhri.2017.11.002. Epub 2018 May 11. PMID 29754016
- [Background] Jonasch E, Donskov F, Iliopoulos O, Rathmell WK, Narayan VK, Maughan BL, Oudard S, Else T, Maranchie JK, Welsh SJ, Thamake S, Park EK, Perini RF, Linehan WM, Srinivasan R; MK-6482-004 Investigators. Belzutifan for Renal Cell Carcinoma in von Hippel-Lindau Disease. N Engl J Med. 2021 Nov 25;385(22):2036-2046. doi: 10.1056/NEJMoa2103425. PMID 34818478
- [Background] Choueiri TK, Bauer TM, Papadopoulos KP, Plimack ER, Merchan JR, McDermott DF, Michaelson MD, Appleman LJ, Thamake S, Perini RF, Zojwalla NJ, Jonasch E. Inhibition of hypoxia-inducible factor-2alpha in renal cell carcinoma with belzutifan: a phase 1 trial and biomarker analysis. Nat Med. 2021 May;27(5):802-805. doi: 10.1038/s41591-021-01324-7. Epub 2021 Apr 22. PMID 33888901
- [Background] Varshney N, Kebede AA, Owusu-Dapaah H, Lather J, Kaushik M, Bhullar JS. A Review of Von Hippel-Lindau Syndrome. J Kidney Cancer VHL. 2017 Aug 2;4(3):20-29. doi: 10.15586/jkcvhl.2017.88. eCollection 2017. PMID 28785532
- [Background] Priesemann M, Davies KM, Perry LA, Drake WM, Chew SL, Monson JP, Savage MO, Johnston LB. Benefits of screening in von Hippel-Lindau disease--comparison of morbidity associated with initial tumours in affected parents and children. Horm Res. 2006;66(1):1-5. doi: 10.1159/000093008. Epub 2006 Apr 27. PMID 16651847
- [Background] Daniels AB, Tirosh A, Huntoon K, Mehta GU, Spiess PE, Friedman DL, Waguespack SG, Kilkelly JE, Rednam S, Pruthi S, Jonasch EA, Baum L, Chahoud J; International VHL Surveillance Guidelines Consortium. Guidelines for surveillance of patients with von Hippel-Lindau disease: Consensus statement of the International VHL Surveillance Guidelines Consortium and VHL Alliance. Cancer. 2023 Oct 1;129(19):2927-2940. doi: 10.1002/cncr.34896. Epub 2023 Jun 19. No abstract available. PMID 37337409
- [Background] Krauss T, Ferrara AM, Links TP, Wellner U, Bancos I, Kvachenyuk A, Villar Gomez de Las Heras K, Yukina MY, Petrov R, Bullivant G, von Duecker L, Jadhav S, Ploeckinger U, Welin S, Schalin-Jantti C, Gimm O, Pfeifer M, Ngeow J, Hasse-Lazar K, Sanso G, Qi X, Ugurlu MU, Diaz RE, Wohllk N, Peczkowska M, Aberle J, Lourenco DM Jr, Pereira MAA, Fragoso MCBV, Hoff AO, Almeida MQ, Violante AHD, Quidute ARP, Zhang Z, Recasens M, Diaz LR, Kunavisarut T, Wannachalee T, Sirinvaravong S, Jonasch E, Grozinsky-Glasberg S, Fraenkel M, Beltsevich D, Egorov VI, Bausch D, Schott M, Tiling N, Pennelli G, Zschiedrich S, Darr R, Ruf J, Denecke T, Link KH, Zovato S, von Dobschuetz E, Yaremchuk S, Amthauer H, Makay O, Patocs A, Walz MK, Huber TB, Seufert J, Hellman P, Kim RH, Kuchinskaya E, Schiavi F, Malinoc A, Reisch N, Jarzab B, Barontini M, Januszewicz A, Shah N, Young WF Jr, Opocher G, Eng C, Neumann HPH, Bausch B. Preventive medicine of von Hippel-Lindau disease-associated pancreatic neuroendocrine tumors. Endocr Relat Cancer. 2018 Sep;25(9):783-793. doi: 10.1530/ERC-18-0100. Epub 2018 May 10. PMID 29748190
- [Background] Dallagnol TN, Da Cas E, Junior OR, Casali-da-Rocha JC. Comprehensive characterization and building of National Registry of von Hippel-Lindau disease in Brazil. Mol Genet Genomic Med. 2023 Apr;11(4):e2136. doi: 10.1002/mgg3.2136. Epub 2023 Jan 10. PMID 36625343
- [Background] Gomy I, Molfetta GA, de Andrade Barreto E, Ferreira CA, Zanette DL, Casali-da-Rocha JC, Silva WA Jr. Clinical and molecular characterization of Brazilian families with von Hippel-Lindau disease: a need for delineating genotype-phenotype correlation. Fam Cancer. 2010 Dec;9(4):635-42. doi: 10.1007/s10689-010-9357-2. PMID 20567917
- [Background] Maher ER, Yates JR, Harries R, Benjamin C, Harris R, Moore AT, Ferguson-Smith MA. Clinical features and natural history of von Hippel-Lindau disease. Q J Med. 1990 Nov;77(283):1151-63. doi: 10.1093/qjmed/77.2.1151. PMID 2274658
- [Background] Kim WY, Kaelin WG. Role of VHL gene mutation in human cancer. J Clin Oncol. 2004 Dec 15;22(24):4991-5004. doi: 10.1200/JCO.2004.05.061. PMID 15611513
- [Background] Rocha JC, Silva RL, Mendonca BB, Marui S, Simpson AJ, Camargo AA. High frequency of novel germline mutations in the VHL gene in the heterogeneous population of Brazil. J Med Genet. 2003 Mar;40(3):e31. doi: 10.1136/jmg.40.3.e31. No abstract available. PMID 12624160
- [Background] Choyke PL, Glenn GM, Walther MM, Patronas NJ, Linehan WM, Zbar B. von Hippel-Lindau disease: genetic, clinical, and imaging features. Radiology. 1995 Mar;194(3):629-42. doi: 10.1148/radiology.194.3.7862955.
- [Background] Chittiboina P, Lonser RR. Von Hippel-Lindau disease. Handb Clin Neurol. 2015;132:139-56. doi: 10.1016/B978-0-444-62702-5.00010-X. PMID 26564077